CLINICAL TRIAL: NCT05613842
Title: Assessment of the Diagnostic Value of 64Cu-SAR-BBN PET Imaging for Men With Negative PSMA PET in Prostate Cancer
Brief Title: Copper-64 SAR Bombesin in PSMA Negative Prostate Cancer (BOP)
Acronym: BOP
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: St Vincent's Hospital, Sydney (Other)
Collaborators: Clarity Pharmaceuticals Ltd (Industry)
Responsible Party: Principal Investigator, Louise Emmett, Professor, St Vincent's Hospital, Sydney
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 062022-01
Record Dates: First submitted 2022-10-31; First posted 2022-11-14 (Actual); Last update posted 2023-09-26 (Actual); Status verified 2023-09

CONDITIONS: Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Intervention Model Description: Male patients 18 years or above with hormone sensitive disease, who demonstrate rising PSA levels (>0.2ng/ml) following definitive therapy and a negative 68Ga-PSMA-11 PET scan (defined as SUV max < 3); Male patients with metastatic castration resistant prostate cancer being considered for 177Lu-PSMA-617 therapy, with known metastatic disease on conventional imaging and sites with low PSMA expression on 68Ga-PSMA-11 PET scan (defined as SUV max <10) in the presence of disease volume of > 1cm.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Male patients with hormone sensitive disease (Experimental): who demonstrate rising PSA levels (>0.2ng/ml) following definitive therapy and a negative 68Ga-PSMA-11 PET scan (defined as SUV max < 3);
  Interventions: Drug: Copper-64 labelled SAR-Bombesin
- Male patients with metastatic castration resistant prostate cancer (Experimental): being considered for 177Lu-PSMA-617 therapy with known metastatic disease on conventional imaging and sites with low PSMA expression on 68Ga-PSMA-11 PET scan (defined as SUV max <10) in the presence of disease volume of > 1cm.
  Interventions: Drug: Copper-64 labelled SAR-Bombesin

INTERVENTIONS:
Drug: Copper-64 labelled SAR-Bombesin — radiolabeled antagonist analog of bombesin for the diagnosis and treatment of gastrin releasing peptide receptor (GRPR)-positive tumors in adults. The product is Copper-64 labelled SAR-Bombesin (Cu-SAR-BBN). Cu-SAR-BBN uses radioactive forms (radionuclide) of copper, copper-64 (64Cu) to image cancers using Positron Emission Tomography (PET) and then copper-67 (67Cu) for therapy by internal beta radiation. 64Cu-SAR-BBN has 3 basic components; the radionuclide (64Cu), bound via MeCOSar (a bifunctional metal chelator, SAR) to a bombesin analog that targets GRPR.
  Other Names: 64Cu-SAR-BBN

SUMMARY:
This phase 2a study will involve enrolment of men presenting with progression of biopsy proven prostate cancer who require imaging for staging/re-staging of their disease. The participants enrolled will be further sub-stratified into two groups; one group of men with hormone-sensitive disease (cohort A), and a second group of men with castrate-resistant disease being considered for 177Lu-PSMA-617 therapy (Cohort B).

DETAILED DESCRIPTION:
This phase 2a study will involve enrolment of men presenting with progression of biopsy proven prostate cancer who require imaging for staging/re-staging of their disease. The participants enrolled will be further sub-stratified into two groups; one group of men with hormone-sensitive disease (cohort A), and a second group of men with castrate-resistant disease being considered for 177Lu-PSMA-617 therapy (Cohort B).

The study will involve men who are being staged or re-staged for metastatic prostate cancer by their treating doctor. The treating doctor will refer the patient to the nuclear medicine department at St. Vincent's Hospital, Sydney for study enrolment.

Screening and D0 visits will be combined for this study. Standard of care bloods (haematology, biochemistry, eGFR and PSA) will be collected at screening/D0 if the results are not already available from the treating doctor. Prior 68Ga-PSMA-11 PET scan within 3 months will be collected from the treating doctor. The PI will ensure that the bloods and 68Ga-PSMA-11 PET scan are reviewed to establish final eligibility before participant undergoes 64Cu-SAR-BBN injection (200mbq) and imaging.

After screening/Day 0 visit, the participant will undergo two imaging scans at 1 hour and 3 hours after having 64Cu-SAR-BBN administration. Total lesional assessment will be calculated with MIM Encore 6.8.7 (MIM Software, Cleveland) using data from the above time points. Safety assessment will be conducted once the participant is enrolled in the study at screening/Day 0 and 48 hours post 3 hours scan by phone call. All adverse events will be recorded on a case report form as source documentation.

ELIGIBILITY:
Inclusion Criteria:

* Ability to provide informed consent documentation indicating that they understand the purpose and procedures required for the study, and are willing to participate in the study;
* Male patients 18 years or above with hormone sensitive disease, who demonstrate rising PSA levels (>0.2ng/ml) following definitive therapy and a negative 68Ga-PSMA-11 PET scan (defined as SUV max < 3);
* Male patients with metastatic castration resistant prostate cancer being considered for 177Lu-PSMA-617 therapy, with known metastatic disease on conventional imaging and sites with low PSMA expression on 68Ga-PSMA-11 PET scan (defined as SUV max <10) in the presence of disease volume of > 1cm.

Exclusion Criteria:

* Significant inter-current acute illness including (but not limited to) requiring the use of intravenous antibiotics, illness associated with any signs of haemodynamic instability, or illness as determined by trial investigators that warrant other emergent treatment;
* ECOG status higher than 2;
* Major surgery (any procedure requiring general anaesthesia) within 6 weeks prior to screening visit;
* History of significant active cancers requiring treatment other than prostate cancer as per Investigator discretion;
* Any other reason that the investigator considers that would make the patient unsuitable to participate in the study.
* eGFR < 40 mL/min/1.73m2

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 30 (Actual)
Dates: Start 2022-08-09 (Actual); Primary Completion 2023-06-06 (Actual); Study Completion 2023-06-06 (Actual)

PRIMARY OUTCOMES:
Explore the diagnostic potential of 64Cu-SAR-BBN PET In men with rising PSA and negative PSMA PET in the 2 cohorts | 24 months
  sensitivity,specificity and accuracy for the detection of primary cancer in %

SECONDARY OUTCOMES:
To assess the diagnostic value of 64Cu-SAR-BBN PET | 24 months
  In the detection of PSMA negative biochemically recurrent or metastatic prostate cancer using a composite standard of truth (biopsy, concurrent imaging and response to targeted therapy)
To evaluate 64Cu-SAR-BBN PET quantitative findings | 24 months
  (SUV max, SUV mean) and sites of metastatic disease and assess the potential for BBN as a therapeutic agent in men with PSMA negative or low PSMA expression disease.
To determine the optimal timing for imaging post BBN injection | 24 months
  with a 1 hour and 3 hours image.

CONTACTS AND LOCATIONS:
Overall Officials: Louise Emmett, Prof, Principal Investigator — Director
Locations (1):
- St Vincent's Hospital, Sydney, New South Wales, Australia

IPD SHARING:
Plan to Share IPD: No